CLINICAL TRIAL: NCT05709704
Title: Comparison of Overall Function Between Postpartum Women With and Without Diastasis Rectus Abdominis
Acronym: DRA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Texas Woman's University (Other)
Collaborators: Wichita State University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-FY2021-405
Record Dates: First submitted 2022-07-07; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Diastasis Recti
Keywords: Overall Function

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postpartum Women WITH DRA: Participants who have the diagnosis of diastasis rectus abdominis
  Interventions: Diagnostic Test: Self-palpation via telehealth; Diagnostic Test: Real-time Ultrasound
- Postpartum Women WITHOUT DRA: Participants who do not have a diagnosis of diastasis rectus abdominis
  Interventions: Diagnostic Test: Self-palpation via telehealth; Diagnostic Test: Real-time Ultrasound

INTERVENTIONS:
Diagnostic Test: Self-palpation via telehealth — This will be used to determine if the participant has the diagnosis
Diagnostic Test: Real-time Ultrasound — This will be used in a subgroup of participants to confirm/rule out a diagnosis

SUMMARY:
The purpose of this research is to examine the effects of diastasis rectus abdominis on the overall function of postpartum women and to determine test-retest reliability and construct validity of a self-assessment palpation of inter-rectus distance for DRA using telehealth.

DETAILED DESCRIPTION:
Step 1: Recruitment

* The investigators will place recruitment fliers in local obstetrician offices, labor and delivery units in local hospitals, retail and daycare establishments, and on social media outlets such as Facebook, Instagram and Twitter.
* The recruitment fliers will ask interested women to email a student investigator to enroll in the research project.

Step 2: Collection of functional outcome data using a Qualtrics version of the Inventory of Functional Status After Childbirth (IFSAC), a demographic survey, a numeric pain reporting scale, Oswestry Low Back Pain Disability Questionnaire, and the Pelvic Floor Distress Index.

Step 3: A meeting time will be set up with every participant to conduct a telehealth visit with a research assistant. During this virtual visit on a private, password protected Zoom call the participant will be instructed on self-assessment palpation of the abdominal wall in order to determine the presence or absence of diastasis rectus abdominis (DRA) along the inter-rectus distance (IRD).

Step 4: The first 18 participants with self-assessed DRA and the first 18 participants without self-assessed DRA, who live in Wichita or surrounding areas, will be scheduled for a one-time in-person confirmation appointment. The appointment will last a maximum of 15 minutes and occur at the WSU Old Town campus room A106. During this confirmation appointment research assistants will screen the participant with the COVID Pre-screening Questions Tool, obtain written informed consent, check the participant in, collect height and weight, and the principal investigator will measure the participants abdominal wall using real-time ultrasound, measure the IRD using the PI's palpation method, and ask the participant to demonstrate and measure IRD using the same palpation method used on the telehealth visit. See the virus protection plan for details of which all participants and investigators will follow in order to minimize risks related to COVID-19).

Step 5: The data will be entered into SPSS and analyzed with appropriate statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18-40 years
* Postpartum (within 6-10 weeks of vaginal delivery)

Exclusion Criteria:

* Women who are currently being treated by a physical therapist for their diastasis rectus abdominis
* Women who had high-risk pregnancies (bedrest, gestational diabetes, pregnancy-induced hypertension)
* Women with a history of abdominal or back surgery
* Women with history of connective tissue disease such as Ehlers-Danlos Syndrome

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The investigators will place recruitment fliers in local obstetrician offices, labor and delivery units in local hospitals, retail and daycare establishments, and on social media outlets such as Facebook, Instagram and Twitter. An announcement will also be included in the Wichita State University Shocker Blast and Strategic Communications. The recruitment fliers will ask interested women to email a research assistant to enroll in the research project.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Inventory of Functional Status after Childbirth | one time between 6-10 weeks postpartum
  Questionnaire used to measure a postpartum woman's ability to function within 5 different domains.

SECONDARY OUTCOMES:
Numeric Pain Scale | one time between 6-10 weeks postpartum
  0-10 scale for the participant to identify any areas of pain in various regions of the body
Oswestry Low Back Pain Disability Index | one time between 6-10 weeks postpartum
  A questionnaire to determine if the participant has any disability in the presence of low back pain
Pelvic Floor Distress Index | one time between 6-10 weeks postpartum
  Questionnaire to determine if the participant has pelvic floor dysfunction

CONTACTS AND LOCATIONS:
Locations (1):
- Wichita State University, Wichita, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided